CLINICAL TRIAL: NCT02113319
Title: An Open-Label, Multicenter, Phase II Study to Assess Dasatinib in Patients With Core Binding Factors Acute Myelogenous Leukemia Refractory to Conventional Chemotherapy or in Molecular Relapse. Intergroupe Français Des leucémie aiguë myéloblastique
Brief Title: Study to Assess Dasatinib in Patients With Core Binding Factors Acute Myelogenous Leukemia
Acronym: DasaCBF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUpromoteur2006-08
Record Dates: First submitted 2014-03-05; First posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2009-01

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Core Binding Factors; Acute Myelogenous Leukemia refractory to conventional chemotherapy; molecular relapse
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dasatinib (Experimental)
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — dasatinib 50 mg and 20 mg During one year

SUMMARY:
In patients with Core Binding Factors Acute Myelogenous Leukemia, the level of Minimal Residual Disease after chemotherapy is predictive of relapse. The relapse risk is also increased in case of mutations of receptors tyrosine kinase. For patients with a high Minimal Residual Disease level at the end of consolidation or in molecular relapse, maintenance by the inhibitor dasatinib is proposed.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting de novo or secondary Core Binding Factors Acute Myelogenous Leukemia
* Patient in first and presenting one of following criteria:
* "Resistant" Patient: decrease of less than 3 log of the Acute Myelogenous Leukemia transcript level in the bone marrow after 2 consolidations
* Patient in " molecular relapse ": increase of of more than 1 log of the Core Acute Myelogenous Leukemia transcript level on two successive marrow samples

Exclusion Criteria:

* Woman of childbearing potential
* Concurrent incurable malignacy other than Acute Myelogenous Leukemia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2007-04; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
measure relapse-free survival | 4 years
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Angers, France